CLINICAL TRIAL: NCT03806699
Title: A Phase 1, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety and Explore the Immunogenicity of ID93+GLA-SE Vaccine in BCG-Vaccinated Healthy Adolescent
Brief Title: Phase 1 Clinical Trial of ID93+GLA-SE Vaccine in BCG-vaccinated Healthy Adolescent
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Quratis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT-QTP101-002
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis, TB, vaccine, adjuvant
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three groups: low dose vaccine, high dose vaccine, or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Since the vials of ID93+GLA-SE and placebo control (normal saline) and their appearances after preparation are different, for double-blinding of the study, the study nurse who administers the study drug or the study pharmacist who stores and manages the study drug will be unblinded to maintain the quality of study blinding. Additionally, an unblinded study monitor will be responsible for confirming the quantity and release of the study drugs. Unblinded study personnels and unblinded study monitor should only be involved in the duties related to administration and/or recording of the study drug, and must not be involved in other duties that may break double-blinding of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Low dose ID93+GLA-SE (Experimental): Participants will receive 0.5 mL (2 μg ID93 + 5 μg GLA-SE) intramuscular injection (IM) into deltoid area, three times in 4-week intervals on Days 0, 28, and 56.
  Interventions: Biological: ID93+GLA-SE
- High dose ID93+GLA-SE (Experimental): Participants will receive 0.5 mL (10 μg ID93 + 5 μg GLA-SE) IM injection into deltoid area, three times in 4-week intervals on Days 0, 28, and 56.
  Interventions: Biological: ID93+GLA-SE
- Control group (Placebo Comparator): Participants will receive 0.5 mL (physiological saline) IM injection into deltoid area, three times on 4-week intervals on Days 0, 28, and 56.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Sterile normal saline
  Arms: Control group
Biological: ID93+GLA-SE — ID93 is a recombinant protein antigen comprising 4 antigens from Mycobacterium tuberculosis (Mtb). The adjuvant GLA-SE is a TLR4 agonist in a stable oil-in-water emulsion.
  Arms: High dose ID93+GLA-SE; Low dose ID93+GLA-SE

SUMMARY:
The purpose of this study is to evaluate safety, immunogenicity of ID93+GLA-SE compared to placebo following three intramuscular (IM) injections on Days 0, 28 and 56 in BCG-vaccinated QFT-negative healthy adolescent. The healthy adolescent will all have had the childhood TB vaccine called BCG, and all of them must have a negative result for a blood test for exposure to the bacteria that cause TB (QuantiFERON-TB Gold Plus, or "QFT"). Study participants will be followed for 12 months after the last injection for safety reasons. Blood will be drawn for laboratory tests for safety and immunogenicity tests. The study hypothesis is that the vaccine is safe and immunogenic in this study population.

DETAILED DESCRIPTION:
After signing a written informed consent to participate in the study(under the premise the legal representative also agree their children participate in the study), subjects will be screened by required assessments per protocol. Eligible subjects who meet the inclusion/exclusion criteria will be randomized in a 1:1:1 ratio to Group 1, Group 2 or Control Group, receiving either ID93+GLA-SE or saline placebo on Days 0, 28 and 56. The investigator will evaluate the safety, immunogenicity of the Investigational Product in the subjects through-out the study.

For safety assessment, subjects will be instructed to record any adverse events in the Subject diary after each vaccination. Subject's safety will be reported to the investigators after 7 days from each vaccination via site visit or a phone call. Solicited AEs will be collected up to 7 days after the final vaccination with the Investigational Product and unsolicited AEs will be collected up to 28 days after the final vaccination with the Investigational Product. For long-term safety assessment of the Investigational Product, serious adverse events and adverse events of special interest will be monitored up to 12 months after the final vaccination with the Investigational Product.

For immunogenicity assessment, blood samples will be collected and analyzed before and after each vaccination. QFT-Gold Plus testing will be performed after 1 month and 12 months from the final vaccination with the Investigational Product.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female who is ≥14 and <19 years of age.
2. History of BCG vaccination that is confirmed through medical examination (i.e., asking a subject about his/her condition) or presence of a scar.
3. Adolescent who are QuantiFERON®-TB Gold Plus negative at screening.
4. Body mass index(BMI) ≥19 and ≤33 (kg/m2) who's Body weight≥40kg at screening.
5. Able to comply with the scheduled visits and are expected to continue working in the current medical institution and be available for a continuous follow-up by the investigator via provided contact information
6. Only for female subjects of childbearing potential:

   * Must be HCG-negative from serum or urine pregnancy test, at screening;

     * Agreed to use one of the following acceptable birth control methods to avoid pregnancy until the end of study (Visit 9): hormonal contraceptives, intrauterine device(IUD) or intrauterine system (IUS), tubal ligation or combination of barrier methods (combined use of barrier methods such as male condoms, female condoms, cervical cap, diaphragm, sponge or implant).
7. Subjects who understand the study procedures and voluntarily decide to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. History of severe chronic disease that may compromise the safety of the subject during the study (e.g., impairment of pulmonary function from tuberculosis infection or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease or uncontrolled epilepsy).
2. Body temperature ≥ 38℃ at the time of randomization or within 24 hours before randomization, from acute fever, acute respiratory diseases, or active infection.
3. Malignant tumors or a history of malignant tumors.
4. Plans to have surgery during the study period.
5. Impaired immune functions including autoimmune disease or immunodeficiency disease.
6. History of Guillain-Barre syndrome.
7. Subjects with a history of anaphylaxis or severe allergic reaction to vaccines, eggs or other allergens.
8. Clinically significant abnormal laboratory values for any of the following tests conducted in the study center, prior to randomization:

   * Hemoglobin, hematocrit, absolute neutrophil count, absolute lymphocyte count or platelet count: < LLN (lower limit of normal)
   * White blood cell count: >ULN (upper limit of normal) or <LLN (lower limit of normal) (i.e., must be within normal limits)
   * ALT, AST, total bilirubin, alkaline phosphatase, creatinine or blood urea nitrogen(BUN): >ULN (upper limit of normal)
9. Received an immunosuppressant, immunity-modifying drug or other treatment that may affect the immune system including cytotoxic anti-cancer agents or radiotherapy, within 3 months before the randomization.
10. Use of systemic steroids (equivalent to daily prednisone ≥ 15mg/day for more than 14 days), inhaled or intranasal steroids, within 3 months before randomization; however, use of topical corticosteroids are acceptable, regardless of dose.
11. Use of immunoglobulin or blood products within 3 months before randomization or plans to use them during the study period.
12. Human Immunodeficiency Virus (HIV) positive at screening.
13. Subjects with chronic hepatitis (e.g., hepatitis B core antibody or hepatitis C antibody positive) at screening.
14. Unable to discontinue current chronic drug therapy such as thyroxin, insulin or other medications with hepatotoxicity or myelotoxicity; however, estrogen and progesterone replacement therapy or contraceptives and topical medications are acceptable.
15. Pregnant or lactating.
16. Use of other vaccines within 4 weeks before screening or plans to use other vaccines from screening to 4 weeks after last IP dosing, plan to use of other vaccines within 4 weeks before End visit.
17. Use of other investigational drugs within 4 weeks before screening.
18. Subjects with history of TB infectivity(Include active, latency TB infection) or positive for Tuberculin Skin Test.
19. Subjects living with a household member who has active TB or infectious TB.
20. Subjects deemed ineligible by investigator based on other reasons.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Solicited AEs for 7 days following each injection, unsolicited AEs for 28 days after each injection, SAEs and AESIs for 12 months after the last injection.
  Solicited (local and systemic reactogenicity), unsolicited (all other adverse events, including laboratory assessments and vital signs), serious AEs and AEs of special interest.

SECONDARY OUTCOMES:
Humoral and cellular immunogenicity assays | Days 0, 28, 56, 84, and 12 months after last injection.
  Immunogenicity will be evaluated by measuring humoral and cellular responses to ID93 + GLA-SE at specified timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hwa Choi, Study Director — Quratis Inc.
Locations (1):
- HALLYM UNIV. Chuncheon Sacred Heart Hospital, Chuncheon, South Korea

IPD SHARING:
Plan to Share IPD: No